CLINICAL TRIAL: NCT06882265
Title: Impact of Remote Vital Signs Monitoring in People Using Long-term Oxygen Therapy : a Randomized Clinical Trial
Brief Title: Impact of Remote Vital Signs Monitoring in People Using Long-term Oxygen Therapy
Acronym: ILD; COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Air Liquide SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 68384723900000068
Record Dates: First submitted 2025-02-18; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-01

CONDITIONS: ILD; COPD
Keywords: Quality of life; Monitoring remote; ILD; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomizations will be carried out blindly, that is, by an evaluator who will not be directly involved in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Monitoring (Experimental): After randomization, participants in the GM group will receive the Venu® SQ monitor (Garmin). All participants will receive guidance on how to use the ODI in the educational class, and at the end they will receive specific instructions for use of the devices they will receive (wearable monitor or pulse oximeter). After the first visit, GM participants will be contacted biweekly by telephone to obtain information on their clinical progress, where they will be asked about the number of exacerbations, respiratory symptoms, medication adherence, time of O2 use, and dyspnea symptoms (mMRC). Likewise, monthly contact will be made to obtain information on health factors associated with quality of life (K-BILD), CAT and EQ-5D-5L, and symptoms of anxiety and depression (HADS).
  Interventions: Behavioral: Group Monitoring
- Control Group (Active Comparator): For the GC, contact will only be monthly to obtain all the information mentioned above in addition to the HR and SpO2 measurements taken on the day of the telephone application.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Group Monitoring — In the intervention group (IG), participants receive a HR and SPO2 monitor watch and a pulse oximeter and will be monitored every 15 days by a nurse to check for non-adherence and/or technical failure, and/or exacerbations, and monthly to apply questionnaires.
  Arms: Group Monitoring
Behavioral: Control Group — In the control group (CG), participants receive only a pulse oximeter and will be monitored monthly by a nurse to administer the questionnaires.
  Arms: Control Group

SUMMARY:
Assess quality of life of patients using prolonged oxygen therapy

DETAILED DESCRIPTION:
Adult participants of both sexes with COPD and PID, prolonged oxygen use, will be evaluated after being informed about the study, agreeing and signing the informed consent form. Participants will be randomized to a control group and a group monitored for 90 days. The monitored group will receive a wearable device to monitor vital signs of heart rate and oxygen saturation and the control group will receive a pulse oximeter. Both groups will be monitored through the cell phone application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical, radiological and/or anatomopathological diagnosis of COPD and ILD according to the 2020 ATS/JRS/ALAT guidelines;
* Age over 18 years;
* Clinical stability (absence of exacerbations or hospitalizations related to the underlying disease) for at least 6 weeks;
* Patients who are on optimized drug therapy, including long-term home oxygen therapy (LTOT)
* Have a smartphone compatible with the monitoring device;
* Signing of the ICF to participate in the study.

Exclusion Criteria:

* Presence of other concomitant lung diseases;
* Myocardial infarction within four months prior to the start of the study, unstable angina or severe heart disease (NYHA functional class III-IV) and/or decompensated.
* Patients who received a lung transplant during the study
* Living outside the coverage area or moving out of state

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life (HRQOL): assessed using the EQ-5D-5L Questionnaire | Change from baseline in 30 days over 90 days
  The EQ-5D-5L questionnaire is a preference-based measure of HRQL with one question for each of five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The responses provided allow for 243 unique health states or can be converted into EQ-5D indices and utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a score ranging from 0 (the worst possible health state) to 100 (the best possible health state).

SECONDARY OUTCOMES:
Clinical Management: The COPD Assessment Test™ (CAT) is a specific questionnaire for COPD that assesses the impact of disease symptoms on quality of life factors in chronic obstructive pulmonary disease. | Change from baseline in 30 days over 90 days
  It consists of eight items related to the health condition and is applied and validated worldwide in several scales. The maximum score for the test is 40 points, and the questions cover the following symptoms: cough, phlegm production, chest pressure, shortness of breath, activities of daily living, psychological aspects, sleep and mood. Each question has six options (0-5), and the lower the score, the better the health condition.
  Time Frame: Change from baseline in 30 days over 90 days
Changes related to quality of life factors in interstitial lung disease - King's Brief Interstitial Lung Disease (K-BILD) | Change from baseline in 30 days over 90 days
  The King's Brief Interstitial Lung Disease (K-BILD) questionnaire is a health status questionnaire developed and validated specifically for patients with ILD. It consists of 15 items that measure health status in the last two weeks in three domains (symptoms, resistance, mental health status and dyspnea on exertion), and is easy to administer and understand by patients. Its classification can range from 0 to 100, with a higher score indicating a higher quality of life, and variations of 5 units are already considered clinically significant.
Change in psychosocial symptoms | Change from baseline in 30 days over 90 days
  Symptoms of anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADs), which consists of 14 items divided into 2 subscales (7 for anxiety and 7 for depression). Each item is scored from 0 to 3, with a maximum score of 21 points for each subscale. A score greater than 8/9 on each subscale suggests a diagnosis of anxiety and/or depression.
Change in dyspnea | Change from baseline in 30 days over 90 days
  Dyspnea scale: modified Medical Research Council (mMRC). The mMRC is a unidirectional 0- to 4-point scale whose questions closely correspond to daily activities that provoke dyspnea.

OTHER OUTCOMES:
Adherence | Baseline
  Evaluated according to the data included in the application and responses to questionnaires.
Exarcebations | Baseline
  Assessed through changes or alterations in vital signs of heart rate and/or oxygen saturation through the wearable
Função pulmonar | Baseline
  Lung volumes will be assessed by spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo (HCFMUSP),, São Paulo, São Paulo, Brazil